CLINICAL TRIAL: NCT06056401
Title: Comparison of Volume-controlled and Pressure-controlled Ventilation in Clasp-knife Position for Robot-assisted Laparoscopic Urological Surgery
Brief Title: Comparison of Volume-controlled and Pressure-controlled Ventilation in Clasp-knife Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Xinyuan, principal investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-FXY-282
Record Dates: First submitted 2023-03-08; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Mechanical Ventilation; General Anesthesia; Urological Surgery; Robotic Surgery
Keywords: Mechanical ventilation; robot-assisted surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCV group (Experimental): For patients assigned in this group, after standard anesthesia, in which the following drugs were used (midazolam 0.05 mg / kg;propofol 1.5-2.5 mg / kg; sufentanil 0.3-0.5 μg / kg; and cisatracurium0.2-0.3 mg / kg), their mechanical ventilation mode was adjusted to the VCV mode.
  Interventions: Behavioral: record Hemodynamic variables, respiratory variables and arterial blood gas at specific times
- PCV group (Experimental): For patients assigned in this group, after standard anesthesia, in which the following drugs were used (midazolam 0.05 mg / kg;propofol 1.5-2.5 mg / kg; sufentanil 0.3-0.5 μg / kg; and cisatracurium0.2-0.3 mg / kg), their mechanical ventilation mode was adjusted to the PCV mode.
  Interventions: Behavioral: record Hemodynamic variables, respiratory variables and arterial blood gas at specific times

INTERVENTIONS:
Behavioral: record Hemodynamic variables, respiratory variables and arterial blood gas at specific times — Hemodynamic variables, respiratory variables and arterial blood gas were measured and recorded 15 minutes after induction of anesthesia (T1), 15 minutes after establishment of a folding knife position (T2), 30 and 60 minutes after CO2 pneumoconiosis (T3 and T4), and 15 minutes after pneumoconiosis (T5). Hemodynamic variables measured included mean arterial pressure , heart rate , cardiac output, cardiac index, stroke volume index and stroke volume variation. Breathing variables include tidal volume, minute ventilation , respiratory rate , airway frontal pressure , mean airway pressure , plateaus airway pressure , peripheral oxygen saturation , oxygen saturation , and oxygen response . Arterial blood gas variables include pH value, arterial carbon dioxide, arterial oxygen pressure , alkali surplus , alveolar oxygen pressure , and bicarbonate of soda ion concentration .

SUMMARY:
Carbon dioxide (CO2) pneumoperitoneum and clasp-knife positioning are commonly used to improve surgical access during robot-assisted laparoscopic urological surgery. However, these methods are sometimes associated with several unwanted cardiopulmonary effects such as increased mean arterial pressure, decreased pulmonary compliance and functional residual capacity, increased peak inspiratory pressure, and respiratory acidosis in association with hypercarbia. Volume-controlled ventilation (VCV) is the most commonly used method of ventilation during general anesthesia. It provides fixed minute ventilation and pulmonary resistance, which affect airway pressure. In pressure-controlled ventilation (PCV), constant inspiratory airway pressure can be achieved by decelerating the flow. However, minute ventilation is not fixed . CO2 pneumoperitoneum in the clasp-knife positioning can influence hemodynamic variables, including blood pressure, heart rate, and cardiac output. This is because changes in airway pressure affect intrathoracic pressure and the function of the heart itself. In this randomized study, we investigated the effects of VCV and PCV on peak inspiratory pressure during robot-assisted laparoscopic urological surgery involving CO2 pneumoperitoneum in the clasp-knife position.

DETAILED DESCRIPTION:
After careful screening, 60 patients were enrolled in the trial. The investigators monitored patients' breathing, circulation and carbon metabolism by measuring arterial gas, cardiac output monitoring, respiratory parameters and circulation parameters at different times in both groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urological surgery in clasp-knife position
* between the age of 18 and 65
* America Society of Anesthesiologist Grades I-II.

Exclusion Criteria:

* Morbid obesity
* systolic blood pressure < 90 mmHg)
* heart rate < 60 beats per minute or > 100 beats per minute
* peripheral blood oxygen saturation < 90%
* Complicated with severe liver and kidney injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Check the patient's ventilation effect at a specific time | T1(15 minutes after induction of anesthesia)
  we recorded the patients' peak inspiratory pressure
Check the patient's ventilation effect at a specific time | T2(15 minutes after position was changed)
  we recorded the patients' peak inspiratory pressure
Check the patient's ventilation effect at a specific time | T3(30 minutes after pneumoperitoneum was established)
  we recorded the patients' peak inspiratory pressure
Check the patient's ventilation effect at a specific time | T4(60 minutes after pneumoperitoneum was established)
  we recorded the patients' peak inspiratory pressure
Check the patient's ventilation effect at a specific time | T5(15 minutes after pneumoperitoneum was released)
  we recorded the patients' peak inspiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Wenqian Lin, Principal Investigator — anesthesiology department of Sun Yat-sen University Cancer Center
Locations (1):
- Cai Xinyuan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No